CLINICAL TRIAL: NCT06912282
Title: Evaluation of Bilateral Single-Electrode VO Combined With STN-DBS Stimulation in the Treatment of Meige Syndrome: A Prospective, Single-Center, Double-Blind, Randomized Controlled Exploratory Clinical Study
Brief Title: Bilateral Single-Electrode VO Combined With STN-DBS for Treating Meige Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jie Hu, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025-084
Record Dates: First submitted 2025-03-26; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Meige Syndrome
Keywords: DBS
MeSH Terms: conditions — Meige Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VO-DBS / VO Combined with STN-DBS Group (Experimental): Patients will undergo bilateral single-electrode VO combined with STN target implantation. After device activation, VO-DBS single-target stimulation will be applied. Evaluation will be conducted after three months, followed by the initiation of combined VO and STN-DBS stimulation.
  Interventions: Device: deep brain stimulation
- STN-DBS / VO Combined with STN-DBS Group (Active Comparator): Patients will undergo bilateral single-electrode VO combined with STN target implantation. After device activation, STN-DBS single-target stimulation will be applied. Evaluation will be conducted after three months, followed by the initiation of combined VO and STN-DBS stimulation.
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation — bilateral single-electrode VO combined with STN target implantation

SUMMARY:
Meige syndrome is a rare and debilitating movement disorder characterized by blepharospasm, oromandibular dystonia, and cervical muscle contractions, often refractory to pharmacological therapies. Deep brain stimulation (DBS), initially developed to treat essential tremor and Parkinson's disease, has been explored in recent years as a potential treatment for various dystonias, including Meige's syndrome. This clinical study aims to evaluate the safety and efficacy of bilateral single-electrode ventralis oralis (VO) nucleus stimulation combined with subthalamic nucleus deep brain stimulation (STN-DBS) in patients with Meige syndrome.

DETAILED DESCRIPTION:
While deep brain stimulation (DBS) targeting the subthalamic nucleus (STN) or the globus pallidus interna (GPi) has shown moderate efficacy, incomplete symptom relief and high stimulation thresholds with associated side effects remain significant limitations. Emerging evidence suggests that dual-target neuromodulation combining STN with ventralis oralis (VO) nucleus stimulation may synergistically modulate hyperactive basal ganglia-thalamocortical circuits, potentially enhancing therapeutic outcomes.The study will involve patients diagnosed with Meige syndrome who are eligible for DBS therapy. Participants will be randomly assigned to one of two groups.The primary outcome measure is the improvement in motor symptoms, assessed using the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) before and after treatment. Secondary outcomes will include changes in quality of life, anxiety and depression scores, and any adverse effects related to the DBS procedure.The results of this study will be used to guide future clinical trials and inform the treatment options for patients with Meige syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the clinical diagnostic criteria for Meige syndrome
* Only includes patients with: Blepharospasm-type Meige syndrome and Blepharospasm with lower jaw muscle dystonia-type
* All patients must have undergone at least one year of systematic and standard treatment prior to surgery

Exclusion Criteria:

* History of neurological diseases other than Meige syndrome
* Severe cognitive impairment
* Severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of primary symptoms | 1 year after stimulation
  Scale title: Burke-Fahn-Marsden Dystonia Rating Scale Section I: Motor subscale (0-120) Section II: Disability scale (0-30) Higher scores: Indicate worse outcomes (more severe dystonia symptoms).

SECONDARY OUTCOMES:
Improvement of symptoms | 1 year after stimulation
  Scale title: Jankovic Rating Scale Minimum value: 0 (No dystonia) Maximum value: 8 (Severe dystonia) Higher scores: Indicate worse outcomes (more severe dystonia symptoms).
Improvement of symptoms | 1 year after stimulation
  Scale title: Blepharospasm Disability Index Minimum value: 0 (No disability) Maximum value: 24 (Severe disability) Higher scores: Indicate worse outcomes (more severe disability due to blepharospasm).
Improvement of symptoms | 1 year after stimulation
  Scale title: Oromandibular Dystonia Questionnaire Minimum value: 0 (No symptoms or disability) Maximum value: 100 (Severe disability) Higher scores: Indicate worse outcomes (more disability due to oromandibular dystonia).
Improvement of symptoms | 1 year after stimulation
  Scale title: Oromandibular Dystonia Rating Scale Minimum value: 0 (No dystonia) Maximum value: 314 (Severe dystonia) Higher scores: Indicate worse outcomes (more severe oromandibular dystonia symptoms).
Psychological assessment | 1 year after stimulation
  Scale title: Hamilton Anxiety Rating Scale Minimum value: 0 (No anxiety) Maximum value: 56 (Severe anxiety) Higher scores: Indicate worse outcomes (more severe anxiety).
Psychological assessment | 1 year after stimulation
  Scale title: Hamilton Depression Rating Scale Minimum value: 0 (No depression) Maximum value: 52 (Severe depression) Higher scores: Indicate worse outcomes (more severe depression).
Cognitive assessment | 1 year after stimulation
  Scale title: Mini-Mental State Examination Minimum value: 0 (Severe cognitive impairment) Maximum value: 30 (No cognitive impairment) Higher scores: Indicate better outcomes (better cognitive function).
Cognitive assessment | 1 year after stimulation
  Scale title: Montreal Cognitive Assessment Minimum value: 0 (Severe cognitive impairment) Maximum value: 30 (No cognitive impairment) Higher scores: Indicate better outcomes (better cognitive function).
health-related quality of life | 1 year after stimulation
  Scale title:Short Form 36 Health Survey
  The SF-36 is a widely used tool to assess general health status and quality of life. It includes 36 items that measure eight health domains:
  Physical functioning Role limitations due to physical health problems Role limitations due to emotional problems Energy/fatigue Emotional well-being Social functioning Pain General health perceptions Each of the domains is scored separately, and the overall score can reflect a person's physical and mental health.
  Minimum value: 0 (Worst health status) Maximum value: 100 (Best health status) Higher scores: Indicate better outcomes (better health-related quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided